CLINICAL TRIAL: NCT00257296
Title: Evaluation of an Intimate Partner Violence Screening-Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Louise-Anne McNutt, Associate Professor, University at Albany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: S1751
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Mass Screening; Methods

ARMS (2):
- Screening and Intervention (Experimental): Use a computer-based screening tool for intimate partner violence and provide a multi-faceted intervention based on the needs of the woman and services should would like to utilize.
  Interventions: Other: Screening and Intervention
- Usual Care (Active Comparator): Use a computer-based screening tool for intimate partner violence and provide list of resources available. Also, all physicians were trained on intimate partner violence and were told they could help anyone regardless of randomization.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Screening and Intervention — Screening for intimate partner violence and providing a multi-faceted intervention which depends on the needs of the patient
  Arms: Screening and Intervention
Other: Usual Care — Screening for intimate partner violence and provide enhanced usual care which includes providing resource list, educating medical staff and partner violence and instructing physicians to help all patients regardless of assigned arm.
  Arms: Usual Care

SUMMARY:
The purpose of the study is to evaluate a multi-faceted intimate partner violence (IPV) screening/intervention targeting abused women who are seen for prenatal care in obstetrics-gynecology clinics or general medical care in internal medicine clinics. The intervention is based on our clinical experience and review of the literature which suggests: 1) IPV can vary and no one pattern exists for all women; 2) recovery from abuse usually occurs over time and not necessarily immediately after it is first detected; 3) women have gone down many different paths leading to an abusive relationship and there is no single path to recovery; 4) for screening/interventions to be credible and ultimately disseminated they must respond to the complexity of the patient stories clinicians see everyday when caring for women experiencing IPV and 5) busy obstetricians/internists/clinicians are unlikely to effectively screen and treat women experiencing IPV unless they are supported by other personnel trained to address IPV as well.

The intervention also is based on recommendations of IPV experts and on the theory of chronic disease management that recognizes that the best outcomes are achieved when: 1) patients are educated and given the support and skills to set their own goals and make their own choices; 2) multidisciplinary teams work better than programs focused only on physician behavior; 3) active monitoring of progress is essential; 4) active coping styles using a range of therapeutic modalities are available and 5) a stepped approach is utilized with those not making progress or with more severe problems receiving the greatest intensity of services.

The screening/intervention will be available to each abused woman for approximately three to six months. Patients in the evaluation study will be surveyed at the following time points: baseline, 1 week, 1 month, 3 months, 6 months, and for the partial cohort that starts early, 9 months. Additionally, a sample of nonabused women will be surveyed at baseline to serve as a referent group.

Our primary hypotheses are, that compared to usual care, abused women receiving the intervention will have a reduction in levels of IPV, decreases in depression and nonspecific physical symptoms, increase in functional health status, increase in safety behaviors, increase in help seeking for issues related to IPV, and reduction of general medical services.

ELIGIBILITY:
Inclusion Criteria:

Females Ages 18 to 45 years Seen at study sites for primary care during study periods Speaks English Able to separate from accompanying person(s) Willing to participant

Exclusion Criteria:

Too ill to participate Unable to separate from accompanying person(s) Unable to speak English Refuse to participant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 471 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2005-10-15 (Actual); Study Completion 2005-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise-Anne McNutt, PhD, Principal Investigator — University at Albany, State University of New York; Daniel Ford, MD, MS, Principal Investigator — Johns Hopkins University